CLINICAL TRIAL: NCT06335121
Title: Implementation of PrEP Care Among Women in Family Planning Clinics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Illinois at Chicago (Other); Planned Parenthood of Illinois (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21120602; 1R01MH134264 (NIH)
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: PrEP Uptake; HIV; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Aim 2 (Experimental): During the intervention period, PPIL staff will capture PrEP eligible women through an updated electronic flag alert in the patient's electronic medical record. The flag will alert to offer the patient PrEP navigation services and implement adapted POWER Up intervention strategies according to training.
  Interventions: Behavioral: POWER Up strategies -
- Control - Aim 2 (No Intervention): PPIL health centers will follow current PrEP navigation procedures using current monitoring system.

INTERVENTIONS:
Behavioral: POWER Up strategies - — Clinics will implement adapted POWER Up intervention strategies when a patient is flagged as PrEP eligible.
  Arms: Intervention - Aim 2

SUMMARY:
This study will evaluate implementation strategies to address barriers and increase uptake of PrEP among Black cisgender women in Planned Parenthood of Illinois (PPIL) health centers.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include ciswomen presenting at a PPIL health center with a positive STI test (syphilis, gonorrhea, or chlamydia) and identified in the EHR using STI testing records and new fields for optimizing support of provider PrEP counseling.

Exclusion Criteria:

- Participants will be excluded if they are not PrEP eligible, have a negative STI test, or are not identified in the EHR.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Ciswomen will be eligible for participation in this study.
Enrollment: 250 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PrEP prescriptions among Black women accessing PPIL services and eligible for PrEP. | 1 month
  PrEP eligibility among Black women will be defined based on positive STI test and identified in the EHR using STI testing records and new fields for optimizing support of provider PrEP counseling. Using de-identified patient-level EHR data for eligible women at each clinic within each time point, we will create a dichotomous variable for having received a prescription for PrEP during a given time period.

SECONDARY OUTCOMES:
Receipt of PrEP refills among Black women accessing FP services at 6 months. | 6 months
  Using de-identified patient-level EHR data for eligible patients at each clinic within each time point, we will create a dichotomous variable for receiving refills of prescriptions for PrEP of those with an initial PrEP prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Haider, MD, MPH, Principal Investigator — Rush University Medical Center; Amy Johnson, PhD, MSW, Principal Investigator — Ann and Robert H. Lurie Children's Hospital of Chicago, Northwestern University Feinberg School of Medicine

IPD SHARING:
Plan to Share IPD: No